CLINICAL TRIAL: NCT03900065
Title: Lappenpräkonditionierung Durch Intermittierende Negative Drucktherapie - Eine Prospektive, Randomisierte, Kontrollierte Klinische Studie
Brief Title: Flap Preconditioning by Intermittent Negative Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Mehran Dadras, MD, Chief resident, Department of Plastic Surgery, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-6408-BR
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Complication of Surgical Procedure; Flap Ischemia
Keywords: flap preconditioning

STUDY DESIGN:
Intervention Model Description: Randomized control trial comparing no preconditioning to preconditioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No preconditioning of the flap.
- Preconditioned group (Experimental): Preconditioning of the flap prior to surgery.
  Interventions: Procedure: Preconditioning

INTERVENTIONS:
Procedure: Preconditioning — Foam-mediated intermittent negative pressure will be applied to the skin of the planned flap for 5 days before surgery.
  Arms: Preconditioned group

SUMMARY:
A randomized controlled trial to investigate the effect of negative pressure preconditioning of flaps on surgical outcome and microcirculation of the tissue.

DETAILED DESCRIPTION:
Flap surgery relies on the perfusion of the transposed or transplanted tissue. Distal parts of flaps are at risk of ischemia leading to wound complications and reoperation. The potential benefit of a preconditioning protocol using foam mediated negative pressure on the flap before surgery is to be examined.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a free or pedicled musculocutaneous M. latissimus dorsi-flap with the time frame of 5 days preconditioning.

Exclusion Criteria:

* Infection of skin of planned flap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of hypoperfused skin island | up to 7 days postoperatively
  The percentage of hypoperfused skin island should be measured clinically after surgery
Skin oxygen saturation of distal flap | 1 day postoperative
  The skin oxygen saturation of distal flap is measured via laserdoppler

SECONDARY OUTCOMES:
Wound complications | up to 12 weeks postoperatively
  wound complications including need of surgical reoperation are assessed
VEGF expression in skin and muscle of flap | once during surgery
  Laboratory examination of tissue specimen obtained during surgery
Density of flap dermal vessels | once during surgery
  Laboratory examination of tissue specimen obtained during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Björn Behr, MD, Principal Investigator — Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil Bochum; Mehran Dadras, MD, Study Director — Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil Bochum
Locations (1):
- Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No